CLINICAL TRIAL: NCT04092075
Title: Safety and Efficacy of the Silk'n Toothbrush (ToothWave), Home Use Device for Reduction of Calculus, Gingivitis and Dental Plaque.
Brief Title: Safety and Efficacy of the ToothWave -12 Weeks Calculus Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DO116551A
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Gingivitis; Plaque; Calculus, Dental
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid; Dental Calculus

STUDY DESIGN:
Intervention Model Description: Single blind prospective study
Who Masked: Outcomes Assessor
Masking Description: The Outcomes Assessors will not be exposed to the type of brush the subject is using or to the group they are assigned to (treatment or control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment group (Experimental): The treatment is conducted with the ToothWave toothbrush Intervention: brushing with Radio frequency (RF)-utilizing powered toothbrush
  Interventions: Device: RF-utilizing powered toothbrush
- Control group (Sham Comparator): Regular powered toothbrush Intervention: brushing with a regular powered toothbrush with no RF
  Interventions: Device: Control placebo with no RF

INTERVENTIONS:
Device: RF-utilizing powered toothbrush — RF-utilizing Powered toothbrush
  Other Names: RF toothbrush
  Arms: Treatment group
Device: Control placebo with no RF — Placebo control, toothbrush with no RF
  Arms: Control group

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the home-use device Silk'n toothbrush (ToothWave) for the improvement in dental health through the reduction of plaque, gingivitis, and calculus.

DETAILED DESCRIPTION:
This is a single blind, prospective study aimed to evaluate the safety and efficacy of the Silk'n toothbrush in reduction of gingivitis, dental plaque and calculus.

The study includes a total of 168 treatment sessions, twice a day, and 5 clinic visits over a period of 12 weeks.

One treatment group (Silk'n toothbrush - ToothWave) and 1 control group (an ADA approved power toothbrush (PTB)) will participate in the study.

For each patient, assessment data will be collected at baseline, 4 weeks, and at 6 weeks. Calculus condition will be measured after 12 weeks in addition to the other timepoints. The average data sets will be calculated for each group.

Treatment is defined as a timed 2 minutes of teeth brushing in a regular manner, twice a day (morning and evening). Brushing will be undertaken using the Silk'n toothbrush and standard fluoride toothpaste. The control group will use a regular PTB and standard fluoride toothpaste.

ELIGIBILITY:
Inclusion Criteria

1. Adult subjects aged 18-70, that are in good health.
2. Subject must have:

   2.1. Baseline gingivitis (MGI) score of at least 1.80. 2.2. Baseline gingival bleeding (GBI) of ≥1 on at least 20 sites. 2.3. Dental Plaque mean score greater than 0.6 according to the RMNPI (Rustogi Modified Navy Plaque Index).

   2.4. Total Calculus deposits greater than 9 according to the Volpe-Manhold Index.
3. Have a minimum of 20 'scorable' teeth (excluding 3rd molars).
4. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects. Subjects will sign the Informed Consent Form.
5. The subjects should be willing to comply with the study procedure and schedule, including the follow up visits.

Exclusion Criteria

1. Current or history of oral cavity cancer or oropharyngeal cancer.
2. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
3. Pregnant or nursing by subject report.
4. Any active condition in the oral cavity at the discretion of the investigator.
5. Any surgery in the oral cavity within 3 months prior to treatment, or before complete healing.
6. Subjects that do not brush regularly.
7. Any condition that might make it unsafe for the subject to participate in this study, at the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Calculus | 12 weeks
  A reduction of calculus deposits as compared to control, as evaluated by Volpe-Manhold Index.

SECONDARY OUTCOMES:
Dental plaque | 6 weeks
  A reduction in the level of dental plaque compared to control, according to Rustogi Modification of the Navy.
Gingival inflammation | 6 weeks
  A reduction in the level of gingival inflammation compared to control, according to the Modified Gingival Index (MGI).

CONTACTS AND LOCATIONS:
Overall Officials: Bennett T Amaechi, BDS, MS, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No